CLINICAL TRIAL: NCT04348539
Title: Evaluation of the Effects of Coordination, Strength and Cardiorespiratory Endurance Training on Physical Fitness, Kinematic and Physiomechanics Parameters of Gait and Indicators Associated With the Quality of Life in Older People
Brief Title: Older People Gait: Physiomechanics and Functionality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Leonardo A. Peyré-Tartaruga, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaitOlderpeople
Record Dates: First submitted 2020-03-25; First posted 2020-04-16 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Old Age; Debility
Keywords: Locomotion; Aging; Training; Physical Fitness; Gait; Quality of life; Health
MeSH Terms: conditions — Frailty | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Balance training (Experimental): The balance training consists of 3 moments: warm up, main and stretch. Warm-up with mobility exercises for major joints and large muscle groups. The main part will have eight exercise stations divided into: a) five balance exercises (dynamic and static with or without object balance) on a varied floor, b) three agility exercises, and a stretching of the worked muscle groups and a final relaxation.
  Interventions: Other: Balance training
- Strength training (Experimental): Muscle strength training will consist of 3 moments: warm up, main and stretch. Warm up with mobility exercises for the main joints and large muscle groups. The main part will include strength exercises with lower and upper limbs with two sets of 6-12 repetitions according to periodization, and a stretching of the muscle groups worked
  Interventions: Other: Balance training
- Cardiorespiratory endurance training (Experimental): The older people walking training consists of 3 moments: warm up, main and stretch. They will do a brief free walking warm-up for 3 minutes in the Self-selected walking speed, then walk according to the training cycle, and then a stretching of the main muscle groups. Will be held, twice a week for 45 minutes each session. The training intensity will follow 60-110% of the volume of the 6-minute Test (6MWT) and the Borg Scale at moderate to difficult intervals. the training
  Interventions: Other: Balance training
- Control group (No Intervention): control group: who will receive educational lectures on health, walking and aging.

INTERVENTIONS:
Other: Balance training — 32 sessions will be held twice a week, with each session taking an average of 45 minutes
  Other Names: Strength training; Cardiorespiratory endurance training
  Arms: Balance training; Cardiorespiratory endurance training; Strength training

SUMMARY:
The aim of study is to investigate gait in active elderly people regarding the kinematic parameters of gait, indicators of physical fitness and quality of life.

DETAILED DESCRIPTION:
Objective: Evaluate and compare the effects of different types of training (balance training, strength training, cardiorespiratory endurance training); in the older people in the variables of physical fitness (dynamic balance, static balance, rate of strength production, flexibility and cardiorespiratory endurance), physiomechanics of gait (length and frequency of stride, time of contact and balance, energy conversion, mechanical work , transport cost, dynamic stability and mechanical efficiency of walking at different speeds), indicators associated with quality of life (depressive symptoms, health-related quality of life, fear of falling). Experimental Design: study experimental randomized. Search Location: Exercise Research Laboratory at the School of Physical Education, Physiotherapy and Dance, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil. Participants: older people from the community of both sexes, aged 60 or over, sedentary. Interventions: In this research, three groups of older people will receive intervention during 4 months of different types of training (balance training, strength training, cardiorespiratory endurance training); and a control group, who will receive educational lectures on health, walking and aging. The training programs will have a duration of 4 months and will be periodized so that the duration of the sessions is same between them. The intensity of the interval training will be manipulated by the subjective effort scale (Borg) and by exercise time. The training programs will have a frequency of two sessions per week and a duration of 45 minutes. In order to evaluate the effects of the training, evaluations will be performed before and after the training period. Outcomes: the results will be related to the variables physical fitness, physiomechanics of gait, and indicators associated with quality of live. Data Analysis: Data will be described by average values and standard deviation values. The comparisons between and within groups will be performed using a Generalized Estimating Equations (GEE) analysis, adopting a level of significance (α) of 0.05, and Bonferroni post-hoc to identify the differences between the means in all variables. Expected Results: The investigators believe that the better the level of physical fitness, the less likely it is that the elderly will enter into a frame of disability or fragility, especially improving physical fitness when compared to the control group. In addition, strategies to protect the elderly can be formulated through physical programs aimed at preventing the functional capacity and quality of life of the elderly. It is expected that the results of the research will be expandable and the possibility of future developments in the scientific, technological, economic, social and environmental.

ELIGIBILITY:
Inclusion Criteria:

* volunteers
* aged over 60 years
* both sexes
* not performing regular physical activity with professional monitoring

Exclusion Criteria:

* not participate in all stages of the evaluation
* severe heart diseases, uncontrolled hypertension, myocardial infarction within a period of less than one year, being a pacemaker;
* stroke or other associated neurological diseases; insanity;
* prostheses in the lower limbs;
* without ambulation conditions.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance | Change from baseline at 16 weeks
  Dynamic balance: Timed Get Up and Go test (distance of 3 meters), which give the time (seconds) that the individual takes to complete the path of the test as fast as possible (without running).
Strength | Change from baseline at 16 weeks
  Lower limb strength: Test to get up and sit on the chair. The individual sits on the chair, with his arms crossed over his chest and at the signal starts the repetitions of getting up and sitting down for a total of 30 seconds. The number of repetitions the subject is able to perform is added.
Cardiorespiratory endurance | Change from baseline at 16 weeks
  cardiorespiratory endurance: 6-minute test. The individual will walk in a 30 meters course for 6 minutes as fast as he can, without running, resulting in the distance covered in that interval.
Static balance | Change from baseline at 16 weeks
  Static balance: force platform by means of the displacement rate of the centre of mass in the anteroposterior (Fx), medium-lateral (Fy) and vertical (Fz) axes. The older people must climb on the platform and unite their feet, keeping their gaze in a fixed linear point, the test will last for 30 seconds, it will be registered with the eyes open and closed

SECONDARY OUTCOMES:
Locomotor Rehabilitation Index | Change from baseline at 16 weeks
  Locomotor Rehabilitation Index: method of determining how close is the self-selected walking speed compared to the Optimum Speed. The results is given in percent, and when Locomotor Rehabilitation Index value is closer to 100 percent, it indicates that the participants are closer to their theoretical optimal walking speed.
Self-selected walking speed | Change from baseline at 16 weeks
  Self-selected walking speed: This outcome will be measure in test of walking treadmill
Anthropometric data - Body mass | Change from baseline at 16 weeks
  Body mass: measure in kilograms before and after interventions.
Depressive symptoms | Change from baseline at 16 weeks
  Geriatric Depression Scale protocol: consists of 15 questions in which participants are asked to answer yes or no in reference to how they felt over the past week (for instance, "Do the patient feel that their life is empty?," Do the patient feel that their situation is hopeless?). Scores range from 0 to 15 with higher scores indicating more depressive symptoms.
Health-related quality of life: Medical Outcomes Study 36 - Item Short Form Health Survey | Change from baseline at 16 weeks
  Medical Outcomes Study 36 - Item Short Form Health Survey: multidimensional questionnaire, formed by 36 items that encompass eight domains (functional capacity, physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health). The maximum score for each domain is 100, with the total sum being a maximum of 150, with zero being "worst" and 150 "best health status".
Fear of falling | Change from baseline at 16 weeks
  Falls Efficacy Scale - International: questions about the concern with the possibility of falling when performing 16 activities, with respective scores from one to four. The total score can vary from 16 (no concern) to 64 (extreme concern).
Anthropometric data - Height | Change from baseline at 16 weeks
  Height: measure in meters before and after interventions.
Anthropometric data - Body Mass Index | Change from baseline at 16 weeks
  Body Mass Index: Weight and height will be combined to report the body mass index in kg/m2.
Spatial Parameter - Stride length | Change from baseline at 16 weeks
  This outcome is measure by stride length in meters.
Temporal Parameter - Swing time, contact time, time of balance | Change from baseline at 16 weeks
  Swing time in seconds, contact time in seconds, time of balance in seconds. The percentage of contact time will be calculated to measure the duty factor in percentual. The swing and contact time in seconds will be aggregated to distance in meters to arrive at frequency (in Hetz).
Parameters of Pendular Mechanism - Internal Work | Change from baseline at 16 weeks
  The transduction between the potential and kinetic mechanical energies of the center of body mass (called the "inverted pendulum" mechanism). The internal work is the mechanical energy fluctuations of the movement of limbs relative to the center of body mass (Wint, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
Parameters of Pendular Mechanism - external work | Change from baseline at 16 weeks
  The transduction between the potential and kinetic mechanical energies of the center of body mass (called the "inverted pendulum" mechanism). The external work is energy fluctuations of the center of body mass with respect to the external environment or surroundings (Wext, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
Parameters of Pendular Mechanism: total mechanical work | Change from baseline at 16 weeks
  The transduction between the potential and kinetic mechanical energies of the center of body mass (called the "inverted pendulum" mechanism). The total mechanical work (Wtot =internal Work + External Work) produced by a body during activity. These outcomes are measured by composite for:(external, internal mechanical work, in Joules).
Parameters of Pendular Mechanism: Recovery | Change from baseline at 16 weeks
  The mechanical energy exchange of the center of mass is quantified by the calculation of the percentage of reconversion of mechanical energy, called Recovery (R), which counts the form that the mechanical energy is saved through the pendulum mechanism of the locomotion. This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.

OTHER OUTCOMES:
Sociodemographic characteristics | Change from baseline at 16 weeks
  Anamnesis with basic information about age, sex, marital status, education, occupation, housing, occurrence of diseases, use of medication.
Cognitive function | Change from baseline at 16 weeks
  Montreal Cognitive Assessment (MoCA), Portuguese version, evaluates 8 domains of cognitive functioning: attention and concentration, executive functions, memory, language, visuoconstructive abilities, conceptual thinking, calculations and guidance. The total score is 30 points; a value = 26 is considered normal.
Lower limb flexibility | Change from baseline at 16 weeks
  Lower limb flexibility: sit and reach test. The individual sits in the chair with his leg extended, slowly leans forward, trying to touch his toes. A measurement is made from the toes to the fingertips.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Alexandre Peyré-Tartaruga, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GONÇALVES, A. K.; et al. Postural balance program: variables related to falls in elderly. Journal of Physical Education, v. 28, 2017